CLINICAL TRIAL: NCT05348993
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Immunogenicity of G03-52-01 in Adult Subjects
Brief Title: Single or Repeat Dose of G03-52-01 in Adult Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: G03-52-01-002
Record Dates: First submitted 2022-03-31; First posted 2022-04-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Healthy; Botulinum Toxin

STUDY DESIGN:
Intervention Model Description: Single dose of G03-52-01 100 mg or placebo or a repeat dose of G03-52-01 (50mg or 100mg) or placebo on days 1 and 45
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized, double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 50 mg dose of G03-52-01 (Experimental): 150 subjects randomized to 50 mg of G03-52-01
  Interventions: Drug: G03-52-01
- 100 mg dose of G03-52-01 (Experimental): 150 subjects randomized to 100 mg of G03-52-01
  Interventions: Drug: G03-52-01
- Placebo (Placebo Comparator): 75 subjects randomized to placebo
  Interventions: Drug: Placebo
- 100 mg dose of G03-52-01 or Placebo (Other): 250 subjects randomized to 100 mg of G03-52-01 or placebo
  Interventions: Drug: G03-52-01; Drug: Placebo

INTERVENTIONS:
Drug: G03-52-01 — G03-52-01 administered intramuscularly
  Arms: 100 mg dose of G03-52-01; 100 mg dose of G03-52-01 or Placebo; 50 mg dose of G03-52-01
Drug: Placebo — placebo
  Arms: 100 mg dose of G03-52-01 or Placebo; Placebo

SUMMARY:
A Phase 2, randomized, double-blind, placebo-controlled single or repeat dose trial

DETAILED DESCRIPTION:
A Phase 2, multicenter, randomized, double-blinded, placebo-controlled study to evaluate a single (100 mg) or repeat dose (50 mg and 100 mg) of G03-52-01 administered by IM injection(s) in adult subjects. Approximately 625 subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent understood and signed prior to screening procedures.
2. Assessed by the Investigator to be a healthy male or healthy, non-pregnant, non-lactating female between the ages of 18 and 65 inclusive on the day of dosing.
3. Able and willing to comply and be available for all protocol procedures and follow-up for the duration of the study.
4. Body Mass Index (BMI) of ≥18.5 and ≤35 kg/m2.
5. Females of child-bearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy test on Day 1 prior to dosing.

   - A woman is considered of childbearing potential unless post-menopausal (≥ 1 year without menses) or surgically sterilized via bilateral oophorectomy, or hysterectomy or bilateral tubal ligation.
6. If the subject is female and of childbearing potential, she agrees to practice abstinence from sexual intercourse with men or use medically effective contraception (methods with a failure rate of < 1% per year when used consistently and correctly) during participation in the study. Acceptable methods include:

   * Hormonal contraception including implants, injections or oral
   * Two barrier methods, e.g., condom and cervical cap (with spermicide) or diaphragm (with spermicide)
   * Intrauterine device (IUD) or intrauterine system
7. Screening clinical laboratory results within normal ranges or are no greater than a Grade 1 and deemed not clinically significant by Medical Monitor (MM) and Principal Investigator (PI). Any subjects with results that are Grade 2 or above according to Appendix B will be excluded.

   - Laboratory values that are outside the range of eligibility but are thought to be due to an acute condition or due to laboratory error may be repeated once.
8. The urine drug screen is negative.

   * For Cohorts 1-3, if a subject has a positive urine drug screen that the PI believes is caused by a currently prescribed medication, (except for THC), the PI may enroll the subject if they meet all inclusion criteria, and none of the exclusion criteria.
   * For Cohort 4, if a subject has a positive urine drug screen that the PI believes is caused by a currently prescribed medication or positive for THC, the PI may enroll the subject if they meet all other inclusion criteria and none of the exclusion criteria.
9. Breathalyzer test is negative.
10. Available for follow-up for the duration of the study.
11. Agrees not to participate in vigorous activity 2 days prior to dosing and 2 days post-dose Day 1 and Day 45 for Cohorts 1-3 and Day 1 for Cohort 4, per Investigator discretion.

Exclusion Criteria:

1. History of a chronic medical condition that would either interfere with the accurate assessment of the objectives of the study or increase the risk profile of the subject.

   - Chronic medical conditions include but are not limited to diabetes; Asthma requiring use of medication in the year before screening; Autoimmune disorder such as lupus, Wegener's, rheumatoid arthritis, thyroid disease; coronary artery disease; chronic hypertension; History of malignancy except low-grade (squamous and basal cell) skin cancer thought to be cured; chronic renal, hepatic, pulmonary, or endocrine disease (except previous asthma which has required no treatment for the past year).
2. Known history of severe allergic reaction of any type to medications, bee stings, food, or environmental factors or hypersensitivity or reaction to immunoglobulins.

   - Severe allergic reactions are defined as any of the following: anaphylaxis, urticaria, or angioedema.
3. Known allergic reactions to any of the study product components present in the formulation or in the processing.
4. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds).
5. Clinically significant abnormal electrocardiogram (ECG) at screening.

   - Clinically significant abnormal ECG results include but are not limited to: complete left or right bundle branch block; other ventricular conduction block except for incomplete RBB; 2nd degree or 3rd degree atrioventricular (AV) block; sustained ventricular arrhythmia; sustained atrial arrhythmia; two Premature Ventricular Contractions in a row; pattern of ST elevation felt consistent with cardiac ischemia; or any condition deemed clinically significant by a study investigator.
6. Positive serology results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies.
7. Febrile illness with temperature ≥38°C within 7 days of dosing. Subjects with acute febrile illness within 7 days of dosing may be rescreened no earlier than 7 days following resolution of symptoms.
8. Female subjects that are pregnant or breastfeeding or intending to become pregnant within the projected duration of the trial starting from the Screening visit until last dose.
9. Donation of blood or blood product within 56 days of enrollment.
10. Is currently participating or has participated in a study with an investigational product (IP) within 28 days preceding Day 1 (documented receipt of placebo in a previous trial would be permissible for trial eligibility)
11. Plans to enroll in another clinical trial that could interfere with safety assessment of the IP at any time during the study period.

    - Includes trials that have a study intervention such as a drug, biologic, or device only
12. Treatment with a mAB within 3 months of Day 1.
13. Receipt of antibody (e.g., tetanus immune globulin [TIG], varicella zoster immune globulin [VZIG], intravenous immunoglobulin [IVIG], IM gamma globulin) or blood transfusion within 6 months or within 5 half-lives of the specific product given.
14. Reported active drug or alcohol or substance abuse/independence or illicit drug use that, in the opinion of the Investigator, would interfere with adherence to study requirements.
15. Use of H1 antihistamines or beta-blockers within 5 days of dosing Day 1 and Day 45 for Cohorts 1-3 and Day 1 for Cohort 4 (PRN use could be allowed with MM approval).
16. Use of any prohibited medication within 28 days prior to study entry or planned use during the study period.

    - Note: Prohibited medications include immunosuppressives (except nonsteroidal anti-inflammatory drugs [NSAIDs]); immune modulators; oral corticosteroids (topical/intranasal steroids are acceptable); anti-neoplastic agents.
17. Previous exposure to botulinum toxin, receipt of antibodies against botulinum toxin, or previous treatment with equine antitoxin.
18. Any previous injection or any planned injection within 4 months after enrollment of botulinum toxin for cosmetic reasons, spastic dysphonia, torticollis, or any other reason.
19. Any illness or condition that in the judgment of the Investigator may affect the safety of the subject or the evaluation of any study endpoint.
20. Is a study site employee, staff, or close relative as defined.

    * PIs and Sub-Investigators
    * Staff who are supervised by the PI, Sub-Investigators
    * Member of the team conducting this clinical trial
    * Children, spouse, partners, siblings, and parents of site staff

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of AEs following administration of G03-52-01 to the final visit (Cohorts 1-3) | 240 Days
  Number of AEs at each visit.
Occurrence of AEs following administration of G03-52-01 to the final visit (Cohort 4) | 120 Days
  Number of AEs at each visit.
Occurrence of SAEs following administration of G03-52-01 to the final visit (Cohorts 1-3) | 240 Days
  Number of SAEs at each visit.
Occurrence of SAEs following administration of G03-52-01 to the final visit (Cohort 4) | 120 Days
  Number of SAEs at each visit.
Occurrence of changes from baseline in PE following administration of G03-52-01 to the final follow-up visit (Cohorts 1-3) | 240 Days
  Number of changes from baselines in PE at each visit.
Occurrence of changes from baseline in PE following administration of G03-52-01 to the final follow-up visit (Cohort 4) | 120 Days
  Number of changes from baselines in PE at each visit.
Occurrence of changes from baseline in vital signs following administration of G03-52-01 to the final follow-up visit (Cohorts 1-3) | 240 Days
  Number of changes from baselines in vital signs at each visit.
Occurrence of changes from baseline in vital signs following administration of G03-52-01 to the final follow-up visit (Cohort 4) | 120 Days
  Number of changes from baselines in vital signs at each visit.
Occurrence of changes from baseline in clinical safety laboratory values following administration of G03-52-01 to the final follow-up visit (Cohorts 1-3) | 240 Days
  Number of changes from baselines in clinical safety labs at visit.
Occurrence of changes from baseline in clinical safety laboratory values following administration of G03-52-01 to the final follow-up visit (Cohort 4) | 120 Days
  Number of changes from baselines in clinical safety labs at visit.
To evaluate the proportion of subjects with target protective concentration (NAC) value > 0.02 U/mL (BoNT/A) or > 0.03 U/mL (BoNT/B) at Day 45 (Cohorts 1-3) | 45 Days
  Number of subjects with target protective concentration (NAC) value > 0.02 U/mL (BoNT/A) or > 0.03 U/mL (BoNT/B) at Day 45
To evaluate the proportion of subjects with target protective concentration (NAC) value > 0.02 U/mL (BoNT/A) or > 0.03 U/mL (BoNT/B) at Day 90 (Cohorts 1-3) | 90 Days
  Number of subjects with target protective concentration (NAC) value > 0.02 U/mL (BoNT/A) or > 0.03 U/mL (BoNT/B) at Day 90
To evaluate the proportion of subjects with target protective concentration (NAC) value > 0.02 U/mL (BoNT/A) or > 0.03 U/mL (BoNT/B) at 4 hours post dose (Cohort 4) | 1 Day
  Number of subjects with target protective concentration (NAC) value > 0.02 U/mL (BoNT/A) or > 0.03 U/mL (BoNT/B) at 4 hours post dose
To evaluate the proportion of subjects with target protective concentration (NAC) value > 0.02 U/mL (BoNT/A) or > 0.03 U/mL (BoNT/B) at 8 hours post dose (Cohort 4) | 1 Day
  Number of subjects with target protective concentration (NAC) value > 0.02 U/mL (BoNT/A) or > 0.03 U/mL (BoNT/B) at 8 hours post dose

SECONDARY OUTCOMES:
To evaluate the proportion of subjects with target protective concentration (NAC) value > 0.02 U/mL (BoNT/A) or > 0.03 U/mL (BoNT/B) at Day 120 (Cohorts 1-3) | 120 Days
  Number of subjects with target protective concentration (NAC) value > 0.02 U/mL (BoNT/A) or > 0.03 U/mL (BoNT/B) at Day 120
To evaluate the proportion of subjects with target protective concentration (NAC) value > 0.02 U/mL (BoNT/A) or > 0.03 U/mL (BoNT/B) at 8 hours post dose (Cohort 4) | 1 Day
  Number of subjects with target protective concentration (NAC) value > 0.02 U/mL (BoNT/A) or > 0.03 U/mL (BoNT/B) at 8 hours post dose
Descriptive statistics of selected PD at all timepoints tested (Cohorts 1-3) | 120 Days
  MNA assessments for BoNT serotypes A and B at pre-dose, 24 hours post dose, and on Days 8, 15, 45 (before repeat-dose), 49, 90, and 120
Descriptive statistics of selected PD at all timepoints tested (Cohort 4) | 90 Days
  MNA assessments for BoNT serotypes A and B at pre-dose, 2 hours, 4 hours, 8 hours, 24 hours and on Days 30, 45, and 90
Descriptive statistics of selected ADA at all timepoints tested (Cohorts 1-3) | 120 Days
  ECLA assessment of ADA titers for each of the mAbs at pre-dose and on Days 90 and 120
Descriptive statistics of selected ADA at all timepoints tested (Cohorts 4) | 240 Days
  ECLA assessment of ADA titers for each of the mAbs at pre-dose and on Days 15, 45 (before repeat-dose or placebo), 60, 90, 120, 150, 180, and 240
Descriptive statistics of selected PK at all timepoints tested (Cohorts 4) | 120 Days
  ELISA/ECLA assessment of AUC(0-t) for each of the mAbs at pre-dose, 2 hour, 4 hours, 8 hours, 24 hours, 72 hours post dose, and on Days 8, 15, 30, 45, 90, and 120

OTHER OUTCOMES:
Descriptive statistics of selected PK parameters at all time points tested of the two lots | 120 Days
  ELISA/ECLA assessment for each of the mAbs at pre-dose, 24 hours, and 72 hours post-dose, and on Days 8, 15, 45 (prior to dosing) 49, 90, and Day 120

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - AMR Mobile, Mobile, Alabama
  - AMR Tempe, Tempe, Arizona
  - AMR Fort Myers, Fort Myers, Florida
  - AMR Miami, Miami, Florida
  - AMR El Dorado, El Dorado, Kansas
  - AMR Newton, Newton, Kansas
  - AMR Wichita West, Wichita, Kansas
  - AMR Wichita East, Wichita, Kansas
  - AMR Lexington, Lexington, Kentucky
  - AMR New Orleans, New Orleans, Louisiana
  - AMR Kansas City, Kansas City, Missouri
  - AMR Las Vegas, Las Vegas, Nevada
  - AMR Norman, Norman, Oklahoma
  - AMR Knoxville West, Knoxville, Tennessee
  - AMR Norfolk, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No